CLINICAL TRIAL: NCT03724136
Title: Alzheimer's Autism and Cognitive Impairment Stem Cell Treatment Study
Acronym: ACIST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MD Stem Cells (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDSC-ACIST
Record Dates: First submitted 2018-10-25; First posted 2018-10-30 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Alzheimer Dementia; Vascular Dementia; Lewy Body Disease; Lewy Body Dementia With Behavioral Disturbance (Disorder); Dementia, Mixed; Parkinson-Dementia Syndrome; Chronic Traumatic Encephalopathy; Huntington's Dementia; Wernicke Korsakoff Syndrome; Traumatic Brain Injury; Dementia, Multi-Infarct; Autism; Autism Spectrum Disorder; Autistic Behavior; Autistic Disorder, Current or Active State; Cadasil; LATE Limbic-predominant Age-related TDP-43 Encephalopathy
Keywords: Dementia; Alzheimer's Disease; CADASIL; Autism Spectrum Disorder; Adult Autism; High Functioning Autism; Asperger's Syndrome; CTE Chronic Traumatic Encephalopathy; TBI Traumatic Brain Injury; LATE Limbic-predominant Age-related TDP-43 Encephalopathy
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Mixed Dementias; Progressive supranuclear palsy atypical; Chronic Traumatic Encephalopathy; Korsakoff Syndrome; Brain Injuries, Traumatic; Dementia, Multi-Infarct; Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive; CADASIL; limbic-predominant age-related TDP-43 encephalopathy; Dementia; Asperger Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of 3 arms with monitoring and retesting at 1,3,6 and 12 months following treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): Intravenous Bone Marrow Stem Cell (BMSC) Fraction
  Interventions: Procedure: Intravenous Bone Marrow Stem Cell (BMSC) Fraction
- Arm 2 (Active Comparator): Intravenous Bone Marrow Stem Cell (BMSC) Fraction combined with Near Infrared Light exposure .
  Interventions: Procedure: Intravenous Bone Marrow Stem Cell (BMSC) Fraction; Procedure: Near Infrared Light
- Arm 3 (Active Comparator): Intravenous Bone Marrow Stem Cell (BMSC) Fraction combined with Intranasal topical Bone Marrow Stem Cell (BMSC) Fraction.
  Interventions: Procedure: Intravenous Bone Marrow Stem Cell (BMSC) Fraction; Procedure: Intranasal Topical Bone Marrow Stem Cell (BMSC) Fraction

INTERVENTIONS:
Procedure: Intravenous Bone Marrow Stem Cell (BMSC) Fraction — 14 cc of BMSC fraction separated from bone marrow aspirate and filtered with 150 micron filter and administered intravenously.
Procedure: Intranasal Topical Bone Marrow Stem Cell (BMSC) Fraction — Approximately 1 cc of BMSC fraction separated from bone marrow aspirate and administered to the nasal mucosa topically.
  Arms: Arm 3
Procedure: Near Infrared Light — Near Infrared Light will be administered using an FDA cleared medical device on the preoperative day and the first postoperative day as tolerated to the general area of the frontal bone.
  Arms: Arm 2

SUMMARY:
The purpose of the study is to evaluate the use of autologous Bone Marrow Derived Stem Cells (BMSC) as a means to improve cognitive impairment as occurs in Alzheimer's Disease and other dementias and to improve behavior and socialization issues which occur in adult Autism Spectrum Disorder. The use of Near Infrared Light, in conjunction with the use of BMSC, will also be assessed.

DETAILED DESCRIPTION:
Cognition is the process of generating thoughts, recalling memories, processing information, and higher order associations including social interactivity that all take place in the brain. It requires sufficient health and interactivity of neurons in the brain including their ability to form and maintain synaptic connections.

Cognitive impairment results from the loss of these abilities. ACIST will test the hypothesis that the delivery of Bone Marrow Derived Stem Cells (BMSC) via the methods in the study with or without the addition of Near Infrared Light will improve cognition through the ability of BMSC to positively affect the health and function of neurons and the brain.

Patients enrolling with cognitive impairment will require assessment with the Mini-Mental Status Exam (MMSE). A score of 24 or less will be required. Progressive dementias such as Alzheimer's Disease (ALZ) show a decline of 2 to 4 points per year on MMSE. The goal for ACIST in progressive and stable dementia will be stability over the 1 year follow up and ideally an improvement of 3 points on MMSE.

Patients enrolling with Autism Spectrum Disorder (ASD) will be required to be adults (over 18 years of age) and to have a score on the Autism Spectrum Quotient of 20 or above. The goal will be a decrease of 5 or more on the scale over the 1 year follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Have documented cognitive impairment or diagnosis of disease associated with cognitive impairment such as Alzheimer's Disease, Autism Spectrum Disorder.
2. If under current medical therapy (pharmacologic or surgical treatment) for the condition be considered stable on that treatment and unlikely to have reversal of the associated cognitive impairment as a result of the ongoing pharmacologic or surgical treatment.
3. In the estimation of the investigator have the potential for improvement with BMSC treatment and be at minimal risk of any potential harm from the procedure.
4. Be over the age of 18
5. Be medically stable and able to be medically cleared by their primary care physician or a licensed primary care practitioner for the procedure. Medical clearance means that in the estimation of the primary care practitioner, the patient can reasonably be expected to undergo the procedure without significant medical risk to health.

Exclusion Criteria:

1. All patients must be capable of an adequate neurologic examination and evaluation to document the pathology.
2. Patients must be capable and willing to undergo follow up neurologic exams with the the investigators or their own neurologists as outlined in the protocol.
3. Patients or their designated responsible party for medical decisions must be capable of providing informed consent. Cognitive or memory impairment does not necessarily mean the patient is incapable of giving informed consent. They may simply need more time to process or repetition of the content of the consent to reach understanding and provide informed consent.
4. In the estimation of the investigator the BMSC collection and treatment will not present a significant risk of harm to the patient's general health or to their neurologic function.
5. Patients who are not medically stable or who may be at significant risk to their health undergoing the procedure will not be eligible.
6. Women of childbearing age must not be pregnant at the time of treatment and should refrain from becoming pregnant for 3 months post treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental Status Exam (MMSE) | 1,3,6 and 12 months post treatment.
  In cognitive impairment patients this standard cognitive function test will be administered. The change from pretreatment baseline to each time point post treatment will be assessed.
Autism Spectrum Quotient Exam | 1,3,6 and 12 months post treatment.
  Patients with Autism Spectrum Disorder (ASD) or Autism will undergo testing with the Autism Spectrum Quotient (AQ) Exam, an autism assessment for adults. The change in scoring from pretreatment baseline to each time point post treatment will be assessed.

SECONDARY OUTCOMES:
Activities of Daily Living | 1,3,6,and 12 months post treatment
  The patients, friends and family will describe changes in abilities to function on a day to day basis.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Levy, MD, Study Chair — MD Stem Cells; Jeffrey Weiss, MD, Principal Investigator — Coral Springs
Locations (3):
- United States (2):
  - MD Stem Cells, Westport, Connecticut
  - MD Stem Cells, Coral Springs, Florida
- Medcare Orthopaedics & Spine Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danielyan L, Schafer R, von Ameln-Mayerhofer A, Buadze M, Geisler J, Klopfer T, Burkhardt U, Proksch B, Verleysdonk S, Ayturan M, Buniatian GH, Gleiter CH, Frey WH 2nd. Intranasal delivery of cells to the brain. Eur J Cell Biol. 2009 Jun;88(6):315-24. doi: 10.1016/j.ejcb.2009.02.001. Epub 2009 Mar 25. PMID 19324456
- [Background] Duncan T, Valenzuela M. Alzheimer's disease, dementia, and stem cell therapy. Stem Cell Res Ther. 2017 May 12;8(1):111. doi: 10.1186/s13287-017-0567-5. PMID 28494803
- [Background] Johnstone DM, Moro C, Stone J, Benabid AL, Mitrofanis J. Turning On Lights to Stop Neurodegeneration: The Potential of Near Infrared Light Therapy in Alzheimer's and Parkinson's Disease. Front Neurosci. 2016 Jan 11;9:500. doi: 10.3389/fnins.2015.00500. eCollection 2015. PMID 26793049
- [Background] Robbins JP, Price J. Human induced pluripotent stem cells as a research tool in Alzheimer's disease. Psychol Med. 2017 Nov;47(15):2587-2592. doi: 10.1017/S0033291717002124. Epub 2017 Aug 14. PMID 28805182
- [Background] Park SE, Lee NK, Na DL, Chang JW. Optimal mesenchymal stem cell delivery routes to enhance neurogenesis for the treatment of Alzheimer's disease: optimal MSCs delivery routes for the treatment of AD. Histol Histopathol. 2018 Jun;33(6):533-541. doi: 10.14670/HH-11-950. Epub 2017 Nov 29. PMID 29185257
- [Background] Shroff G. Human Embryonic Stem Cells in the Treatment of Autism: A Case Series. Innov Clin Neurosci. 2017 Apr 1;14(3-4):12-16. eCollection 2017 Mar-Apr. PMID 28584692
- [Background] Chez M, Lepage C, Parise C, Dang-Chu A, Hankins A, Carroll M. Safety and Observations from a Placebo-Controlled, Crossover Study to Assess Use of Autologous Umbilical Cord Blood Stem Cells to Improve Symptoms in Children with Autism. Stem Cells Transl Med. 2018 Apr;7(4):333-341. doi: 10.1002/sctm.17-0042. Epub 2018 Feb 6. PMID 29405603
- [Background] Weiss JN, Levy S. Neurologic Stem Cell Treatment Study (NEST) using bone marrow derived stem cells for the treatment of neurological disorders and injuries: study protocol for a nonrandomized efficacy trial. Clin Trials Degener Dis. 2016 [cited 2019 Jun 18];1:176-80.
- See also: Report from CNN on Duke University stem cell autism study — https://www.cnn.com/2017/04/05/health/autism-cord-blood-stem-cells-duke-study/index.html